CLINICAL TRIAL: NCT02252523
Title: Feasibility of Dexmedetomidine-based Sedation in Neurocritical Care Patients : a Pilot Study
Brief Title: Dexmedetomidine-based Sedation in Neurocritical Care Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-210; 2013-004697-10 (EudraCT Number)
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Acute Brain Injuries
Keywords: Feasibility study
MeSH Terms: conditions — Brain Injuries | interventions — Dexmedetomidine

ARMS (1):
- DEXMEDETOMIDINE (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
This will be an open, prospective pilot study with pharmacological analysis. This study is designed to assess the efficacity and safety of dexmedetomidine-based sedation in two subgroups of neurocritically ill patients requiring mechanical ventilation for more than 48 hours. Those with or at risk for intracranial hypertension requiring deep sedation and those requiring a light to moderate sedation for early neurological evaluation.

The main objective is to assess the feasability of dexmedetomidine infusion in terms of efficacy and safety (especially cardiovascular tolerance) in brain-injured patients admitted to intensive care unit and requiring sedation and mechanical ventilation for a predictable duration greater than or equal to 48 hours. Secondary objectives include the study of hemodynamic parameters evolution, dose-response relationship, blood (+/- cerebrospinal fluid) drug concentration, opioates and co-hypnotic consumption.

DETAILED DESCRIPTION:
A written informed consent will be obtained from patients next-of-kin, before study enrollment according to inclusion and exclusion criterias. All consecutive brain-injured patients (traumatic brain injury, subarachnoid or intracerebral hemorrhage, postoperative neurosurgical procedure) admitted to our neurocritical care unit, older than 18 years and requiring sedation and analgesia for mechanical ventilation longer than 48 hours, will be eligible for the study. Depending on the absence or presence of lesion which may increase intracranial pressure, patients will be included in the "light to moderate" sedation subgroup (MLS) or in the "deep" sedation subgroup (DS).

In the MLS subgroup (RASS 0/-3), sedation and analgesia will be drived by propofol and opiates. Once the goals of sedation achieved with usual hypnotic, dexmedetomidine will be initiated at a dose of 0.5 μg/kg/h, and then gradually increased or decreased by increments of 0.1 μ g / kg / h all hours to a maximum dose of 1.4 μg/kg/h, depending on the target sedation achievement. Propofol will be discontinued at study drug initiation. Dexmedetomidine infusion will bemaintained at least during 48 hours, evaluation of the efficacy and safety will be continuous during this period.

After these first 48 hours, in the absence of neurological worsening requiring a deep sedation and if sedation's levels will are achieved with dexmedetomidine alone (ie without requirement of propofol continuous administration) , it will be maintained untill withdrawal of mechanical ventilation. Otherwise, study drug will discontinued and propofol will be restarted.

In the DS subgroup, "deep" sedation (RASS -4/-5) will be achieved by propofol infusion. If sedation level are not achieved with the maximum recommended propofol dose (5mg/kg/h), midazolam will be started to reach target sedation level with a maximum dose of 0.15mg/kg/h. Once the goals of sedation will be achieved a dexmedetomidine infusion will be initiated at a dose of 0.5 μg/kg/h and then gradually titrated by increase of 0.1 μg/kg/h every hour up to the maximum patient-tolerated dose (maximum dose of 1.4 μg/kg/h). Conventional hypnotic doses will be adjusted according to the sedation target. In parallel to dexmedetomidine titration, midazolam first and then propofol will be decreased. The study drug will be maintained at the maximum patient-tolerated dose for a total of 48 hours during which the efficacy and safety will be assessed continuously. After this period, dexmedetomidine will be discontinued. According to the patient's neurological evolution, either sedation objectives will remain identical (RASS -4/-5), or sedation will be decreased. Conventional hypnotic will be used again to achieve these objectives.

The expected result of this study is to confirm that the administration of dexmedetomidine is effective and safe for "light to moderate" and "deep" sedation of brain-injured patients admitted to intensive care unit. In addition, this feasibility study could provide legitimacy if the results are conclusive, to conduct a prospective multicenter randomized controlled trial on the potential benefits of dexmedetomidine in neurocritical ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Brain-injured patients (traumatic brain injury, subarachnoid or intracerebral hemorrhage, postoperative neurosurgical procedure)
* Older than 18 years
* Requiring sedation and analgesia for mechanical ventilation longer than 48 hours
* Written informed consent obtained from patients next-of-kin, before study enrollment
* Depending on the absence or presence of lesion which may increase intracranial pressure, patients will be included in the "light to moderate" sedation subgroup or in the "deep" sedation subgroup

Exclusion Criteria:

* - Heart rate < 45 bpm,
* Uncontrolled shock or cardiac failure,
* High-grade AV block,
* Acute ischemic neurological injury,
* Severe liver failure,
* Drug overdose and prior enrollment in a trial with any experimental drug in the last 30 days,
* Need for ongoing neuromuscular blockade except for tracheal intubation,
* Pregnancy/lactation,
* Known allergic reaction to dexmedetomidine,
* Uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic events | at day 1
Adverse effects other than hemodynamic event | at day 1
Premature discontinuation of dexmedetomidine infusion | at day 1
Delirium assessed by CAM- ICU scale | at day 1
Withdrawal syndrome at dexmedetomidine discontinuation | at day 1

SECONDARY OUTCOMES:
Level of sedation assessed by the RASS scale from dexmedetomidine initation | at day 1
Dose of dexmedetomidine necessary to achieve the objectives of sedation | at day 1
Effective plasma concentration | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France